CLINICAL TRIAL: NCT01220687
Title: Administration of Inhaled Nitric Oxide (iNO) as an Adjunct to Neonatal Resuscitation Protocol: A Pilot Trial
Brief Title: Inhaled Nitric Oxide (iNO) as an Adjunct to Neonatal Resuscitation
Acronym: iNO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1976
Record Dates: First submitted 2010-10-07; First posted 2010-10-14 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Respiratory Distress Syndrome in Premature Infants; Very Low Birth Weight Baby
Keywords: Prematurity; Oxygen exposure; Nitric Oxide
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants; Premature Birth | interventions — Nitrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo 20ppm (Placebo Comparator): Nitrogen at 20 ppm at the beginning of study start with gradual taper at 10 minutes of the study and completely off by 17 minutes of the study
  Interventions: Other: Nitrogen
- Inhaled Nitric Oxide (iNO) 20 ppm (Experimental): Inhaled Nitric Oxide 20 ppm at the beginning of study start with gradual taper at 10 minutes of the study and completely off by 17 minutes of the study
  Interventions: Drug: iNO

INTERVENTIONS:
Drug: iNO — Immediately after birth, subjects will be randomized to receive iNO (20ppm) or nitrogen (placebo gas) with blended oxygen (starting with 0.3). Fraction of inspired oxygen will be adjusted by 0.1 increments every 15 seconds targeting pre-ductal oxygen saturation of 70-85% in the first 2 minutes of life, and then 85-93% until the end of the study period while requiring supplemental oxygen.
  Other Names: Inhaled Nitric Oxide
  Arms: Inhaled Nitric Oxide (iNO) 20 ppm
Other: Nitrogen — Subjects will be randomized to receive iNO (20ppm) or nitrogen (placebo gas) with blended oxygen (starting with 0.3). Fraction of inspired oxygen will be adjusted by 0.1 increments every 15 seconds targeting pre-ductal oxygen saturation of 70-85% in the first 2 minutes of life, and then 85-93% until the end of the study period while requiring supplemental oxygen.
  Arms: Placebo 20ppm

SUMMARY:
This study hopes to determine whether nitric oxide along with oxygen during the first 20 minutes of life in infants needing help with breathing will reduce the percentage and total exposure to oxygen during that time frame. Although the use of oxygen in management of breathing is an important part of supporting baby immediately after delivery, there is more evidence that too much exposure to oxygen may lead to potential problems for your baby later. Oxygen exposure can be harmful to premature babies developing lungs.

DETAILED DESCRIPTION:
Current Neonatal Resuscitation Program (NRP) guidelines suggest the use of supplemental oxygen up to fraction of inspired oxygen of 1.0 during neonatal resuscitation for both term and preterm newborns. Exposure to supplemental oxygen in preterm babies has been shown to have significant toxicity. Even minimal exposure in the first hours of life has been shown to be associated with morbidity including later onset of cancer. The transition from fetal circulation to neonatal circulation is a complex process requiring lung inflation and decrease in pulmonary vascular resistance. Endogenous nitric oxide, along with oxygen, plays a major role in facilitating this transition by decreasing pulmonary vascular resistance. It is not known whether exogenous nitric oxide would facilitate this transition. In this study, we propose a novel approach to resuscitation of preterm infants where inhaled nitric oxide (iNO) will be used as an adjunct to oxygen with the primary goal of reducing supplemental oxygen exposure. This study is designed to be a double-blind, randomized, -placebo- controlled pilot trial with strict monitoring of parameters during transition in the delivery room.

ELIGIBILITY:
Inclusion Criteria:

* Infants that are 25 0/7 - 31 6/7 weeks gestation
* Infants who require Continuous Positive Airway Pressure (CPAP) or Positive Pressure Ventilation ( PPV) during delivery room resuscitation.

Exclusion Criteria:

* Refusal of consent
* Known complex congenital anomalies of the heart or lungs
* Known major genetic defects
* Hydrops fetalis

Ages: 1 Minute to 2 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2011-04; Primary Completion 2017-01 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kris Sekar, M.D., Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Oklahoma, Childrens Hospital, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No
Abstract presented to The Pediatric Academic Society Meeting, May 9, 2017

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women admitted in preterm labor with gestational ages of 25 0/7 to 31 6/7 weeks gestation were approached for prenatal consent. 171 mothers were identified, 95 mothers consented
Pre-assignment Details: 64 consented mothers or infants met subsequent exclusion criteria. Of those, only 33 were enrolled at time of delivery. Most common exclusion was aging out of gestational age limit, precipitous delivery, or no team available.
Groups:
- iNO 20 Ppm: Nitric Oxide 20 ppm at the beginning of study start with gradual taper at 10 minutes of the study and completely off by 17 minutes of the study
  iNO: Immediately after birth, subjects will be randomized to receive iNO (20ppm) or nitrogen (placebo gas) with blended oxygen (starting with 0.3). Fraction of inspired oxygen will be adjusted by 0.1 increments every 15 seconds targeting pre-ductal oxygen saturation of 70-85% in the first 2 minutes of life, and then 85-93% until the end of the study period while requiring supplemental oxygen.
Period: Overall Study
Arm/Group | Placebo 20ppm | iNO 20 Ppm
Started | 16 | 15
Completed | 14 | 14
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo 20ppm | iNO 20 Ppm | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: Weeks] — Gestational Age at birth in Weeks
  Weeks | 28.1 [26.7 to 29.1] | 28.6 [27 to 29.9] | 28.4 [26.7 to 29.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 7 | 11 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10 | 10 | 20
  African American | 1 | 1 | 2
  Native American | 1 | 2 | 3
  Hispanic | 2 | 0 | 2
  Other Race | 0 | 1 | 1
Birthweight [Median (Inter-Quartile Range); unit: Grams] | 1105 [780.9 to 1336.9] | 1145 [670 to 1282.5] | 1105 [735.25 to 1277.5]
Apgar Score at one minute [Median (Inter-Quartile Range); unit: units on a scale] — Scale of 0-10 with 0 indicating no heart rate, no respirations, unresponsive to 10 vigorous, pink, active, good heart rate and respirations.
  units on a scale | 5 [4 to 7] | 4 [2 to 5] | 4 [2.25 to 7]
Apgar Score at 5 minutes [Median (Inter-Quartile Range); unit: units on a scale] — Scale of 0-10 with 0 indicating no heart rate, no respirations, unresponsive to 10 vigorous, pink, active, good heart rate and respirations.
  units on a scale | 8 [7 to 8] | 7 [6 to 8] | 7.5 [6.25 to 8]
Any Antenatal Steroid [Count of Participants; unit: Participants] | 8 | 9 | 17
Chorioamnionitis [Count of Participants; unit: Participants] | 2 | 3 | 5
Rupture of Membranes (ROM) greater than 18 hours [Count of Participants; unit: Participants] | 2 | 4 | 6
Maternal Preeclampsia [Count of Participants; unit: Participants] | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Maximum Factional Inspired Oxygen Percent (FiO2)
Description: To investigate whether iNO decreases the supplemental oxygen exposure in the preterm infants who require continuous positive airway pressure (CPAP) or positive pressure ventilation (PPV) during resuscitation as per Neonatal Resuscitation Program (NRP) protocol.
Time Frame: 20 minutes
Measure: Mean (Inter-Quartile Range); unit: percentage of Inspired Oxygen
Arm/Group | Placebo 20ppm | iNO 20 Ppm
Number analyzed (Participants) | 14 | 14
percentage of Inspired Oxygen | 48 [34.73 to 68.20] | 39 [20.98 to 53.26]
Statistical Analysis 1: Comparison: Placebo 20ppm vs iNO 20 Ppm; Test type: Superiority; p = 0.0012, t-test, 2 sided; Mean Difference (Final Values) = 9

2. Primary Outcome: Rate of Hyperoxia
Description: FiO2 >60% at any 5 second increment during the study period of 20 minutes for each infant in each arm.
Time Frame: 20 minutes
Measure: Number; unit: Observations on >60% FiO2
Arm/Group | Placebo 20ppm | iNO 20 Ppm
Number analyzed (Participants) | 14 | 14
Observations on >60% FiO2 | 708 | 370
Statistical Analysis 1: Comparison: Placebo 20ppm vs iNO 20 Ppm; Test type: Superiority; p < 0.0001, Poisson; Rate Ratio = 1.91, 95% CI 2-sided [1.68 to 2.18]

3. Primary Outcome: Pre and Postductal Saturation Levels
Description: Oxygen saturations as described as preductal (right hand) as well as post ductal (either foot) and measured as percent of saturated hemoglobin by pulse oximetry.
Time Frame: at 20 minutes (end of study)
Measure: Mean (Standard Deviation); unit: Percent Saturation
Arm/Group | Placebo 20ppm | iNO 20 Ppm
Number analyzed (Participants) | 14 | 14
Percent Saturation
  Preductal Saturation | 90.5 (5.7) | 82.8 (13.8)
  Postductal Saturation | 79.9 (25.8) | 78.2 (20)

4. Primary Outcome: Heart Rate During Resuscitation
Description: Measured and recorded heart rates every 5 seconds on study as described as beats per minute (BPM)
Time Frame: 5, 10 and 20 minutes on study
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | Placebo 20ppm | iNO 20 Ppm
Number analyzed (Participants) | 14 | 14
BPM
  BPM at 5 minutes | 139 (53) | 130 (46)
  BPM at 10 minutes | 161 (53) | 149 (46)
  BPM at 20 minutes | 168 (53) | 158 (46)

5. Primary Outcome: Need for Intubation
Description: Infants requiring placement of endotracheal tube as part of the Neonatal Resuscitation Program algorithm for airway management.
Time Frame: by end of study, 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 20ppm | iNO 20 Ppm
Number analyzed (Participants) | 14 | 14
Participants | 4 | 4

6. Secondary Outcome: Intraventricular Hemorrhage > Grade 2
Description: Intraventricular Hemorrhage (IVH) > Gr 2 as described by radiographic scale as described in "Incidence and evolution of subependymal and intraventricular hemorrhage: a study of infants with birth weights less than 1,500 gm.", Papile L A; Burstein J; Burstein R; Koffler H, The Journal of pediatrics, (1978 Apr) Vol. 92, No. 4, pp. 529-34. Journal code: 0375410. ISSN: 0022-3476. L-ISSN: 0022-3476.
  IVH classification systems Papile system Grade I Subependymal hemorrhage Grade II IVH without ventricular dilation Grade III IVH with ventricular dilation Grade IV Extensive IVH with parenchymal involvement
Time Frame: Hospital Discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 20ppm | iNO 20 Ppm
Number analyzed (Participants) | 14 | 14
Participants | 2 | 0

7. Secondary Outcome: Infants With Patent Ductus Arteriosus (PDA) Requiring Treatment
Description: Count of patients requiring either pharmacologic or surgical treatment for persistent PDA
Time Frame: Prior to infant discharge from the hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 20ppm | iNO 20 Ppm
Number analyzed (Participants) | 14 | 14
Participants | 4 | 1

8. Secondary Outcome: Retinopathy of Prematurity (ROP)> Stage 2
Description: Staging of any retinal disease as described by the standard screening by the American Association for Pediatric Ophthalmology and Strabismus. Only infants who survived to obtain retinal imaging are included (12 in Placebo arm and 11 in INO arm)
Time Frame: Prior to infant discharge from the hospital
Population: 2 of the 14 patients in the placebo arm died and had no ROP exam, 3 of the 14 patients in the INO Group died and had no ROP exam.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 20ppm | iNO 20 Ppm
Number analyzed (Participants) | 12 | 11
Participants | 4 | 1

9. Secondary Outcome: Mechanical Ventilation, Non-invasive Ventilation (NIV), and Length of Stay in Days (LOS)
Description: endotracheal or other airway placement and mechanical ventilation in days, days of non-invasive ventilation as described as nasal ventilation, CPAP, high flow and low flow oxygen as counted in days. Only infants who survived to discharge were included in this analysis.
Time Frame: Prior to infant discharge from the hospital
Population: 2 of the 14 patients in the placebo arm died were not included in the analysis, 1 of the 14 patients in the INO Group was excluded for pulmonary hypoplasia..
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo 20ppm | iNO 20 Ppm
Number analyzed (Participants) | 12 | 13
Days
  Mechanical Ventilation | 14 [2 to 29] | 8.5 [1.5 to 26]
  NIV | 15 [3 to 23] | 20.5 [6.5 to 31]
  LOS | 52 [48 to 88] | 70.5 [49 to 108.5]

10. Secondary Outcome: Bronchopulmonary Dysplasia
Description: Bronchopulmonary Dysplasia as described as oxygen need at 36 weeks adjusted gestational age. Only infants who survived to 36 weeks gestation were included in this analysis.
Time Frame: at 36 weeks adjusted gestational age of participant
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 20ppm | iNO 20 Ppm
Number analyzed (Participants) | 12 | 13
Participants | 5 | 5

11. Secondary Outcome: Late Onset Sepsis
Description: Late Onset Sepsis as described as infection after day 5 of life. This would include all patients who survived to day of life 5.
Time Frame: at any time during study period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 20ppm | iNO 20 Ppm
Number analyzed (Participants) | 13 | 12
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded until discharge from the hospital, average age at discharge for all infants who completed study.
Arm/Group | Placebo 20ppm | iNO 20 Ppm
All-Cause Mortality (participants affected / at risk) | 1/14 | 2/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

LIMITATIONS AND CAVEATS:
Small sample size. Recruitment was terminated before reaching our initial target sample size due to precipitous and emergent deliveries, unavailability of the team or baby ineligible due to gestational age at birth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No